CLINICAL TRIAL: NCT04552301
Title: Assessing Inflammatory and Behavioral Pathways Linking PTSD to Increased Asthma Morbidity in WTC Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Juan Wisnivesky, Chief of Division of General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 16-0945
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Asthma; PTSD
Keywords: World Trade Center; Cognitive Processing Therapy; Asthma; Intervention; Pilot Randomized Control Trial
MeSH Terms: conditions — Asthma; Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Data from the observational component of the study will be used to identify WTC workers with asthma and PTSD for the pilot. Eligibility will be determined based on Asthma Control Questionnaire (ACQ) score >1.5, indicating uncontrolled asthma and results of the Structured Clinical Interview for DSM-5 Disorders (SCID) and/or PCL-5 showing evidence of PTSD. Participants will be consented by trained research staff and randomized 1:1 (stratified by level of asthma control) into an intervention (combined asthma self-management and cognitive processing therapy for PTSD) or an active attention control arm (supportive psychotherapy plus asthma education) after completing their 12-month visit.
Who Masked: Outcomes Assessor
Masking Description: Research coordinators (RCs) are blinded to study randomization and treatment arm for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy and Targeted Asthma Education (Experimental): Intervention group - Cognitive Processing Therapy and Targeted Asthma Education
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Targeted Asthma Education
- Psychotherapy and General Asthma Education (Active Comparator): Control group - Psychotherapy and General Asthma Education
  Interventions: Behavioral: Psychotherapy; Behavioral: General Asthma Education

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Integrated CPT. CPT is based on a social cognitive theory of PTSD that focuses on how the traumatic event is construed and coped with by a person who is trying to regain a sense of mastery and control in his or her life. The asthma components that will be integrated into the intervention include psychoeducation about asthma, barriers to asthma self-care, asthma medication education, inhaler technique, and asthma self-management behaviors.
  Other Names: CPT
  Arms: Cognitive Processing Therapy and Targeted Asthma Education
Behavioral: Psychotherapy — The Study Interventionist will conduct generalized supportive psychotherapy with the participants to provide emotional support for both PTSD and general education for asthma.
  Arms: Psychotherapy and General Asthma Education
Behavioral: Targeted Asthma Education — The manualized 10-session program of asthma self-management
  Other Names: Asthma Education
  Arms: Cognitive Processing Therapy and Targeted Asthma Education
Behavioral: General Asthma Education — A 10-session program of similar time
  Other Names: Asthma Education
  Arms: Psychotherapy and General Asthma Education

SUMMARY:
Asthma and post-traumatic stress disorder (PTSD) are the most common conditions in World Trade Center (WTC) rescue and recovery workers. In this study, the study team will evaluate the interplay of biological and behavioral mechanisms explaining the relationship of PTSD with increase asthma morbidity and adapt and pilot test a novel intervention to improve outcomes of WTC workers.

DETAILED DESCRIPTION:
SIGINIFICANCE: Importance of the Problem: Multiple studies have shown a high prevalence of asthma in WTC rescue and recovery workers, local residents, and passersby. Using data from the National Health Interview Survey (NHIS), the researchers found that WTC workers have twice the risk of asthma compared to the general United States (US) population. Data from the WTCHP shows a 28% cumulative incidence of asthma 9 years after September 11, 2001 among WTC workers. These studies show that asthma is the most prevalent respiratory condition among WTC rescue and recovery workers.

WTC workers with asthma include individuals with prior history of the disease and new cases of irritant-induced asthma. Many workers with preexistent asthma developed worsening symptoms after WTC-related exposures (WTC-exacerbated asthma). Other workers developed new asthma symptoms without latency during or after WTC exposure and were diagnosed with irritant-induced asthma. Multiple cases of new onset asthma among WTC workers have been reported in the years following exposure to the WTC site; characterization of these cases has been more difficult. Despite this potential heterogeneity, these conditions are frequently grouped in clinical practice as WTC-related asthma and managed similarly.

Studies found substantial burden of asthma morbidity in WTC workers and exposed community members, with reports of poorly-controlled in 34% and very poorly-controlled symptoms in 35% of exposed individuals. Increased risk of emergency department (ED) visits and hospitalizations as well as poor quality of life in WTC workers with asthma have been reported, showing a major impact on health.

Scientific Premise of Project: PTSD is Associated with Increased Asthma Morbidity in WTC Workers: Prevalence of psychological symptoms in WTC-exposed populations is high; with PTSD reported as the most common (~30%) mental health condition. Studies have also found high rates (25-35%) of PTSD comorbidity in WTC workers with asthma. Mental health conditions and PTSD in particular, have been associated with increased asthma morbidity. The researchers found that WTC workers with PTSD had worse asthma control, increased healthcare use, and poorer quality of life (see preliminary data). Similarly, a study of WTC workers indicated that severity of PTSD symptoms predicted new onset and worsening of asthma. Data from studies in the general population have also shown that PTSD is associated with higher asthma morbidity. In summary, studies have documented a high level of overlap between asthma and PTSD in WTC workers and other exposed populations and have documented that PTSD is a major contributor to increased asthma morbidity. However, the underlying mechanisms explaining this relationship remain unknown.

Potential Biological Pathways Linking PTSD and Asthma Morbidity: The impact of PTSD extends to multiple organ systems as a consequence of changes in the hypothalamic-pituitary axis, the autonomic nervous system, and the immune system.These PTSD-associated systemic alterations may impact asthma morbidity. PTSD is associated with a basal low-grade systemic inflammation, in particular, increased plasma levels of pro-inflammatory cytokines such as interleukin (IL)-1α, IL-2, IL-6, tumor necrosis factor-alpha (TNF-α and decreased IL-4, IL-5 ("Th2-cytokines"). Airway inflammation, a central feature of asthma, may be modulated by enhanced systemic inflammation as that observed in PTSD. Major asthma endotypes, which describe asthma subtypes based on inflammatory mechanisms, include allergic, intrinsic (non-atopic), and noneosinophilic asthma. Allergic asthma is characterized by airway eosinophilia driven by TH2-dominant inflammation. Noneosinophilic asthma is characterized by airway neutrophilia has been associated with refractory disease, severe exacerbations, and increased risk of intubation. Key cytokines driving neutrophilic asthma include IL-1β, IL-6 and IL-17, which are elevated in patients with PTSD.51 IL-6 directs and stabilized T-cells towards a Th17 subset, which can then recruit and activate of neutrophils. Therefore, systemic inflammatory changes associated with PTSD, may worsen asthma outcomes by driving a neutrophilic asthma phenotype. Identification of the biological pathways underlying worse asthma in patients with comorbid PTSD has important implications for disease management including indications for inhaled corticosteroids (ICS) and new biological drugs and may offer new alternative targets for therapy.

Symptom Perception in Asthma Patients with Comorbid PTSD: Effective asthma SMB requires the patient to recognize and respond (use of rescue medication, contact physician, etc.) to their symptoms. Self-monitoring of symptoms is also key for assessing response to treatment and thus, developing effective self-regulatory mechanisms (i.e., ICS linked to improved symptoms; see theoretical framework). Unfortunately, the symptoms that asthma patients experience do not always align with objective measures of their airway obstruction. Experiments have identified 3 asthma symptom perception phenotypes that have important clinical implications: symptom under-perceivers, normal perceivers, and over-perceivers. Prior studies have shown a strong relationship between misperception of symptoms and increased asthma morbidity.

While PTSD is associated with increased objective and subjective asthma morbidity markers, the associations with subjective measures are stronger. The researchers found that PTSD had strong associations with disease control measures and quality of life in WTC workers with asthma. However, the association with FEV1 was weaker (see preliminary data). Other studies had similar findings. These data strongly suggest that over-perception of symptoms may be prevalent among WTC workers with PTSD and may contribute to increased asthma morbidity and complicate SMB. The hypotheses for over-perception of symptoms among WTC workers with PTSD is based on Janssens's cognitive-affective model of symptom perception. A central factor in this model is negative affect common among patients with PTSD. Janssens's model89 proposes that negative affect will be linked with over-perception of symptoms via an associative learning mechanism. Because asthma exacerbations cause a negative affective state, an association between such a state and asthma symptoms develops in patients with PTSD. As a consequence, subsequent negative emotional states due to PTSD may results in the report of severe asthma symptoms in the presence of mild or no airway obstruction. The effect of negative affect is most pronounced on the affective component (i.e., unpleasantness dimension) of dyspnea. Thus, PTSD patients may perceive more asthma symptoms due to perceptions of unpleasant sensations of dyspnea.

PTSD is also characterized by a disruption in the ability to regulate emotions, which can lead to exaggerated emotional reactions to asthma-symptoms, in turn leading to symptom magnification. One relevant cognitive vulnerability factor common to PTSD and asthma is anxiety sensitivity, the tendency to catastrophically misinterpret the bodily sensations associated with anxious arousal (e.g., shortness of breath or chest pounding) as threatening. Anxiety sensitivity is more common among patients with asthma, strongly implicated in the experience of dyspnea, and associated with poor asthma control, and greater behavioral avoidance. Recent work by Dr. Gonzalez (Consultant) indicates that anxiety sensitivity, physical concerns in particular, plays a significant role in understanding the PTSD-asthma symptom link in WTC workers (see preliminary data).

Assessing Asthma Symptom Perception: Symptom perception is typically measured in laboratories by self-reported respiratory symptoms while inducing airway constriction with histamine or methacholine. However, this approach produces biased data because it generates anxiety and primes patients for certain reactions. In contrast, measurements in naturalistic settings (e.g., their home), as the researchers propose to do, is a validated method that reduces the emotional threat of the test environment and omits pharmacological techniques and devices that may generate anxiety.

PTSD May Negatively Impact Asthma SMB: Asthma self-management encompasses several complex behaviors such as adherence to controller medications, adequate inhaler technique, use of action plans, allergen avoidance, and avoiding tobacco exposure that are critical for adequate disease control. Adherence to controller medications in particular, is a factor that heavily influences the outcomes of asthmatics. Studies conducted in the general population and the preliminary data from WTC workers shown that only ~50% of patients with asthma adhere to controller therapy or other SMB.

Mental health conditions are associated with low adherence to chronic disease SMB. PTSD, in particular, has been strongly associated with low treatment adherence in multiple chronic diseases.With smoking being an important part of asthma self-management, it is of special concern that higher rates of smoking have been reported among WTC workers with PTSD. Thus, low adherence to SMB may mediate, in part, the association between PTSD and increased asthma morbidity. However, there is limited data regarding the relationship between PTSD and asthma SMB in the general population or among WTC workers, in particular.

Theoretical Framework: Pathways Mediating the Influence of PTSD on SMB: The researchers will use the Self-regulation Model (SRM) to guide the exploration of the relationship between PTSD and asthma SMB via illness beliefs, emotional representations and symptoms perception. According to the SRM, people with chronic illness, like asthma, compare their somatic sensations (i.e., symptoms) to their "normal" self, and interpret deviations from "normal" in relation to their mental model of their illness, which in turn guides their SMB. Appraisal of the efficacy of their actions (i.e., improved asthma control) serves as a feedback loop to reinforce or modify SMB. The SRM posits five domains of cognitive representations of illness: identity (disease labels), cause (etiology and triggers), timeline (chronicity), consequences (perceived impact), and control (extent to which an illness can be controlled). For example, if asthma patients accurately perceive their respiratory symptoms (identity) and believe asthma is persistent (timeline) they will engage in SMB. The SRM also predicts that patients will be adherent if they learn, via feedback loops, that their asthma medications can prevent symptoms (controllability). Emotional responses to asthma (i.e., worry, upset, or anxious) also influence SMB. The framework of the SRM is highly useful for identifying the modifiable beliefs and emotional mechanisms which underlie behaviors worth targeting for self-management support interventions. The researchers expect that PTSD may impact asthma SMB in several ways. WTC workers with PTSD may magnify asthma symptoms (identity) when they are actually experiencing negative emotions. Over-perception of symptoms could be a major barrier for internalizing positive feedback loops about medication effectiveness, leading to low adherence. WTC workers with PTSD and asthma may also misinterpret the causes of their asthma symptoms and thus, avoid situations that trigger the physical sensations they fear. Paradoxically, decreasing the frequency of PTSD symptoms via avoidance of perceived (not actual) asthma triggers may contribute to illness representations that focus more on this maladaptive avoidance, and less on SMB. Some patients view asthma as a chronic (timeline) inflammatory condition (cause), which requires adherence to daily ICS. Data from non-WTC asthma populations shows that patients with PTSD are more likely to view asthma as an acute, episodic disease.This 'acute' representation of asthma has been associated to low medication adherence. Patients with PTSD also tend to feel out of control (due to unexpected symptoms and catastrophic thoughts) and have lower self-efficacy, which has been linked to low ICS adherence. According to the SRM, emotional responses also influence SMB. As discussed above, patients with PTSD have emotional regulation difficulties; thus, strong negative emotional reactions to asthma may deplete WTC workers' self-regulatory resources managing emotions to the detriment of asthma SMB.SRM has also shown that medication beliefs strongly predict ICS adherence. Negative affect in workers with PTSD may extend to patients' beliefs about ICS (e.g., side effects, dependence, etc.) negatively influencing adherence. Moreover, patients with PTSD may avoid asthma medications and awareness of symptoms because these factors may serve as trauma cues or reminders of 9/11, triggering memories of their WTC traumatic experiences. Thus, this copying style (avoidance) may lead to low medication adherence.

Absence of Interventions Integrating PTSD and Asthma Management: Despite the strong link between asthma and PTSD in WTC workers, there are no interventions aimed at managing both conditions. Dr. Gonzalez is conducting a randomized clinical trial (RCT) to evaluate an integrative mind-body treatment, the 3RP, to improve the management of PTSD and lower respiratory symptoms in WTC workers (see preliminary data). The 3RP is an 8-session group-based program that seeks to promote the physiological, emotional, cognitive and behavioral effects of the relaxation response.The 3RP program focuses on 3 major areas to decrease stress and build resiliency: 1) eliciting the relaxation response via sustained mental focus with an attitude of open receptive awareness; 2) promoting stress awareness and decreasing reactivity, which involves identification of the 5 components of one's stress response (thoughts, emotions, physical reactions, behaviors, and relationship changes) and learning skills (e.g., cognitive restructuring) to change these components; and 3) increasing use of adaptive strategies by focusing on skills to promote positive growth and self-efficacy in response to stress. However, this intervention was not specifically developed for WTC workers with asthma and thus, does not address misperception of symptoms or disease SMB.

ELIGIBILITY:
Inclusion Criteria:

- Pilot inclusion criteria:

* Diagnosed with PTSD based on SCID or PCL-5
* Poorly controlled asthma based on ACQ score ≥1.5; and
* Completion of observational study 12-month visit.

Exclusion Criteria:

* Active Suicidal Ideation
* Co-existence of COPD or other chronic respiratory illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Wisnivesky, MD, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wisnivesky JP, Becker JH, Ankam J, Markowitz SB, Doernberg M, Dickens B, Busse P, Crowley L, Federman A, Katz C, Weiss JJ, Gonzalez A. The Relationship Between Post-Traumatic Stress Disorder and Self-Management Behaviors in World Trade Center Workers with Asthma. J Allergy Clin Immunol Pract. 2022 Jan;10(1):242-249. doi: 10.1016/j.jaip.2021.08.035. Epub 2021 Sep 14. PMID 34534721
- [Background] Wisnivesky JP, Markowitz SB, James S, Stone K, Dickens B, Busse P, Crowley L, Federman A, Katz C, Gonzalez A. Comorbid posttraumatic stress disorder and major depressive disorder are associated with asthma morbidity among World Trade Center workers. Ann Allergy Asthma Immunol. 2021 Mar;126(3):278-283. doi: 10.1016/j.anai.2020.10.007. Epub 2020 Oct 22. PMID 33098982
- [Background] Wisnivesky JP, Agrawal N, Ankam J, Gonzalez A, Busse P, Lin J, Federman A, Feldman J, Weiss JJ, Markowitz SB. World Trade Center workers with asthma and post-traumatic stress disorder perceive airflow limitation more accurately. Ann Allergy Asthma Immunol. 2024 Jan;132(1):62-68. doi: 10.1016/j.anai.2023.08.005. Epub 2023 Aug 12. PMID 37580015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants did not have their baseline demographic info because they were added later on in the pilot study
Groups:
- Psychotherapy and General Asthma Education: Psychotherapy and General Asthma Education
  Psychotherapy: The Study Interventionist will conduct generalized supportive psychotherapy with the participants to provide emotional support for both PTSD and general education for asthma.
  General Asthma Education: A 10-session program of similar time
Period: Overall Study
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 participants did not have their baseline demographic info because they were added later on in the pilot study
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (7.7) | 51.9 (8.3) | 54.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White or Caucasian | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported or Other | 2 | 2 | 4
  Hispanic or Latino | 2 | 8 | 10
Education [Count of Participants; unit: Participants]
  8th grade or less | 0 | 0 | 0
  Some high school | 0 | 2 | 2
  High school or GED | 2 | 3 | 5
  1 to 3 years of college | 7 | 8 | 15
  4-year college graduate | 2 | 1 | 3
  Higher degree | 0 | 2 | 2
  Missing information | 1 | 0 | 1
Monthly income [Count of Participants; unit: Participants]
  Less than $3000 | 6 | 8 | 14
  More than $3000 | 6 | 7 | 13
  Missing Information | 0 | 1 | 1
Marital status [Count of Participants; unit: Participants]
  Unmarried | 9 | 5 | 14
  Married | 3 | 11 | 14
Language [Count of Participants; unit: Participants]
  Mostly English | 11 | 10 | 21
  Mostly Spanish | 1 | 4 | 5
  About the same | 0 | 2 | 2
Smoking status [Count of Participants; unit: Participants]
  Current/former smoker | 4 | 3 | 7
  Never smoker | 6 | 12 | 18
  Missing Information | 2 | 1 | 3
Insurance [Count of Participants; unit: Participants]
  Medicare | 4 | 3 | 7
  Medicaid | 2 | 3 | 5
  Medicare and Medicaid | 1 | 1 | 2
  Private | 3 | 7 | 10
  Other | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5), is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Full range from 0-80, higher score indicates more symptoms.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 39.2 (10.3) | 36.4 (9.6)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 32.9 (14.7) | 34.3 (11.3)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 29.8 (17.4) | 30.9 (9.1)

2. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: The ACQ assess asthma beliefs about asthma control. The ACQ is a 7-item instrument, full scale from 0-6, higher score indicates more impairment.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 2.1 (1.1) | 2.1 (0.4)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 1.7 (1.0) | 2.0 (2.1)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 1.9 (1.5) | 2.1 (0.9)

3. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: The AQLQ assess asthma beliefs about asthma quality of life. The AQLQ is a 32-item instrument, full scale from 1-7, higher score indicates better health outcomes
Time Frame: Baseline, 1 week post-intervention, 3 months post-intervention
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 3.7 (1.1) | 3.7 (0.8)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 4.3 (1.2) | 3.9 (1.0)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 4.4 (1.6) | 3.8 (1.0)

4. Secondary Outcome: Medication Adherence Report Scale (MARS)
Description: The MARS assess asthma beliefs about asthma medication adherence. The MARS is a 10-item instrument, full range from 0-10, higher score indicates higher likelihood of medication adherence.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 4.4 (0.8) | 4.5 (0.7)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 4.5 (0.6) | 4.5 (1.1)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 4.6 (0.6) | 4.5 (0.8)

5. Secondary Outcome: Illness Perception Questionnaire (IPQ)
Description: The IPQ assess asthma beliefs about illness perception. The IPQ is an 80-item instrument, total scale from 0-80, with higher score indicating higher perception of effects on illness.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 47.0 (14.3) | 46.8 (12.3)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 41.4 (10.3) | 44.0 (12.3)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 42.7 (13.1) | 44.6 (12.9)

6. Secondary Outcome: Beliefs About Medicines Questionnaire (BMQ)
Description: Beliefs About Medicines Questionnaire (BMQ), a 10-item validated tool assessing medication necessity and concerns. The BMQ consists of two five-item scales assessing patients' beliefs about the necessity of medication and their concerns about taking it. Each item scored on a five-point Likert scale, ranging from 1 = strongly disagree to 5 = strongly agree. Total subscale scores for the Necessity and Concerns Scales range from 5 to 25. Higher scores indicate stronger beliefs.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention Necessity Score | 20.1 (2.8) | 19.5 (3.2)
  1 Week Post-Intervention Necessity Score: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention Necessity Score | 20.7 (1.8) | 19.4 (4.1)
  3 Months Post-Intervention Necessity Score: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention Necessity Score | 19.5 (3.5) | 18.8 (3.7)
  Pilot Baseline Pre-Intervention Concerns Score | 16.3 (2.7) | 17.2 (4.0)
  1 Week Post-Intervention Concerns Score: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention Concerns Score | 16.0 (3.7) | 16.9 (4.4)
  3 Months Post-Intervention Concerns Score: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention Concerns Score | 17.1 (4.6) | 16.0 (4.3)

7. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) Depression Severity
Description: As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 12.9 (5.4) | 10.9 (4.9)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 9.7 (4.6) | 10.4 (6.4)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 10.1 (7.5) | 9.7 (5.8)

8. Secondary Outcome: Generalized Anxiety Disorder-7
Description: The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
  Full scale from 0-21, with higher score indicating poorer health outcomes.
Time Frame: Baseline; 1 week post-intervention, up to 11 weeks; 3 months post-intervention, up to 5.5 months
Population: Data available for participants who completed instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
Number analyzed (Participants) | 19 | 19
score on a scale
  Pilot Baseline Pre-Intervention | 11.1 (5.1) | 9.4 (4.6)
  1 Week Post-Intervention: number analyzed (Participants) | 10 | 14
  1 Week Post-Intervention | 10.1 (5.6) | 8.9 (5.7)
  3 Months Post-Intervention: number analyzed (Participants) | 11 | 15
  3 Months Post-Intervention | 9.3 (7.8) | 8.1 (5.2)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Cognitive Processing Therapy and Targeted Asthma Education | Psychotherapy and General Asthma Education
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT04552301/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04552301/ICF_001.pdf